CLINICAL TRIAL: NCT01147575
Title: Effects of Creatine Supplementation in Rett Syndrome: A Randomized, Placebo-controlled Trial
Brief Title: Effects of Creatine Supplementation in Rett Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: M Freilinger, MD, Medical University Vienna, Department of Pediatric and Adolescent Medicine
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: OENB11758
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-05

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome, Randomized, Methylation
MeSH Terms: conditions — Rett Syndrome | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creatine monohydrate (Active Comparator): The patients received orally 200 mg CMH per kg body weight divided in three doses per day. Following period 1 (6 months) of supplementation and a wash-out period of 4 weeks without CMH respectively the groups were switched for another 6 months (period 2).
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): The patients received orally 200 mg Placebo per kg body weight divided in three doses per day in identically prepared capsules. Following period 1 (6 months) of supplementation and a wash-out period of 4 weeks without Placebo respectively the groups were switched for another 6 months (period 2).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — The patients received orally 200 mg CMH per kg body weight divided in three doses per day. Following period 1 (6 months) of supplementation and a wash-out period of 4 weeks without CMH the groups were switched for another 6 months (period 2).
  Arms: Creatine monohydrate
Dietary Supplement: Placebo — The patients received orally 200 mg Placebo per kg body weight divided in three doses per day. Following period 1 (6 months) of supplementation and a wash-out period of 4 weeks without placebo the groups were switched for another 6 months (period 2).
  Arms: Placebo

SUMMARY:
Creatine supplementation in RTT: a randomized controlled trial

Rett Syndrome (RTT) is a neurodevelopmental disorder characterised by apparently normal early development (stage 1 of RTT) followed by loss of purposeful hand use, distinctive hand stereotypes, slow brain growth, loss of language, respiratory irregularities, gastrointestinal disturbances, gait abnormalities, seizures, and mental retardation. These symptoms typically appear between 6 and 18 months of age (stage 2). Subsequently, there is gradual stabilisation of severe mental retardation and motor compromise (stage 3). The majority (70% to 80%) of patients show mutations in the methyl-CpG-binding-protein-2 (MeCP2) gene, located on chromosome Xq28. MeCP2 encodes a transcription repressor protein that is ubiquitously expressed in all tissues.

As RTT primarily affects females, only very few males with mutations in MeCP2 have been identified. Mutations in MeCP2 have also been identified in children with X-linked mental retardation, autism and a clinical phenotype that resembles Angelman Syndrome.

The aim of this study is to investigate the effects of a dietary supplement on the biochemical and clinical parameter of RTT. About 80 % of labile methyl groups generated through the re-methylation cycle are used for the synthesis of creatine within the human organism. Supplementation of creatine will therefore increase the availability of labile methyl groups for different methylation reactions including methylation of DNA.

The study will be double blind and cross-over. The patients will get creatine monophosphate (200 mg/kg/d in three dosages per day) or placebo. After 6 months and a wash-out period of 4 weeks the groups are changed for the next 6 months.

All participants with RTT and mutations in MeCP2 will undergo physical and neurological exam, quantitative EEG, behavioral assessment, laboratory testing, and neuropsychological evaluations. Participants will have a follow-up after 3, 6, 10, 13 and 16 months (3 months after finishing the study), which will include similar assessments.

ELIGIBILITY:
Inclusion Criteria:

* RTT Syndrome, diagnosed by current consensus criteria

Exclusion Criteria:

* taking supplements containing either folic acid or vitamin B12 or knowingly consuming any vitamin-fortified food items

Ages: 3 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Global DNA Methylation in serum | 6 months
  Global DNA methylation as one primary outcome measure is analyzed at time 0 and after 6 months.
Rett Syndrome Motor and Behavioral Assessment (RSMBA) | 6 months

SECONDARY OUTCOMES:
Metabolic markers of methylation cycle | 6 months
  Markers: Methionine (µmol/l), Homocysteine (µmol/l), SAM (µmol/l), SAH (µmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Freilinger, MD, Principal Investigator — Medical University Vienna, Dep. Pediatrics
Locations (1):
- Medical University Vienna, Dep. of Pediatric and Adolescent Medicine, Vienna, Austria

REFERENCES:
- [Derived] Freilinger M, Dunkler D, Lanator I, Item CB, Muhl A, Fowler B, Bodamer OA. Effects of creatine supplementation in Rett syndrome: a randomized, placebo-controlled trial. J Dev Behav Pediatr. 2011 Jul-Aug;32(6):454-60. doi: 10.1097/DBP.0b013e31822177a8. PMID 21654506